CLINICAL TRIAL: NCT01833988
Title: The Summer Camp Study: Feasibility of Outpatient Automated Blood Glucose Control With a Bi-Hormonal Bionic Endocrine Pancreas in a Pediatric Population at the Clara Barton Diabetes Camps
Brief Title: The Summer Camp Study: Blood Glucose Control With a Bi-Hormonal Bionic Endocrine Pancreas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Boston University (Other)
Responsible Party: Principal Investigator, Steven J. Russell, MD, PhD, Assistant Professor of Medicine, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2013p000561
Record Dates: First submitted 2013-04-13; First posted 2013-04-17 (Estimated); Results first posted 2017-08-11 (Actual); Last update posted 2017-09-08 (Actual); Status verified 2017-08

CONDITIONS: Type 1 Diabetes
Keywords: bionic pancreas; artificial pancreas; insulin; glucagon; continuous glucose monitoring (CGM); outpatient; insulin pump; pediatrics; children; camp; summer camp
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance; Muscle Cramp

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bi-hormonal Bionic Pancreas (Experimental): Bi-hormonal Bionic Pancreas
  Interventions: Device: Bi-hormonal Bionic Pancreas
- Usual Care (Active Comparator): Usual Care
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: Bi-hormonal Bionic Pancreas — Automated blood glucose control via a closed-loop bionic pancreas device.
  Other Names: Boston University Bionic Pancreas
  Arms: Bi-hormonal Bionic Pancreas
Other: Usual Care — Comparator week to closed-loop control, utilizing usual camp care and the subject's own insulin pump.
  Arms: Usual Care

SUMMARY:
This study will test the hypothesis that a wearable automated bionic pancreas system that automatically delivers both insulin and glucagon can improved glycemic control vs. usual care for young people with type 1 diabetes 12-20 in a diabetes camp environment.

DETAILED DESCRIPTION:
The bionic pancreas will be compared to usual care in a crossover design in which each volunteer will serve as his or her own control. Each volunteer will be under closed-loop glucose control for five days and usual camp level of diabetes care for five days in random order with a one day washout period in between.

ELIGIBILITY:
Inclusion Criteria:

* Age 12-20 years with type 1 diabetes for at least one year.
* Diabetes managed using an insulin infusion pump and rapid- or very-rapid-acting insulins including insulin aspart (NovoLog), insulin lispro (Humalog), and insulin glulisine (Apidra) for at least three months prior to enrollment.
* Otherwise healthy (mild chronic disease such as asthma will be allowed if well controlled that do not require medications that result in exclusion).

Exclusion Criteria:

* Unable to provide informed assent
* Unable to comply with study procedures.
* Current participation in another diabetes-related clinical trial other than one that is primarily observational in nature.
* Total daily dose (TDD) of insulin that is > 2 units/kg.
* Pregnancy (positive urine HCG), plan to become pregnant in the immediate future, or sexually active without use of contraception
* Hypoglycemia unawareness (self-reported or legal guardian report of consistent lack of hypoglycemia symptoms when BG is < 50 mg/dl)
* End stage renal disease on dialysis (hemodialysis or peritoneal dialysis).
* History of prolonged QT or arrhythmia
* History of congenital heart disease or current known cardiac disease
* Acute illness (other than non-vomiting viral illness) or exacerbation of chronic illness other than type 1 diabetes at the time of the study.
* Seizure disorder or history of hypoglycemic seizures or coma in the last five years
* Untreated or inadequately treated mental illness (indicators would include symptoms such as psychosis, hallucinations, mania, and any psychiatric hospitalization in the last year), or treatment with second generation anti-psychotic medications, which are known to affect glucose regulation.
* Electrically powered implants (e.g. cochlear implants, neurostimulators) that might be susceptible to radiofrequency interference.
* Use non-insulin, injectable (e.g. exenatide, pramlintide) or oral (e.g. thiazolidinediones, biguanides, sulfonylureas, meglitinides, dipeptidyl peptidase-4 inhibitors, acarbose)anti-diabetic medications.
* History of adverse reaction to glucagon (including allergy) besides nausea and vomiting.
* Unwilling or unable to completely avoid acetaminophen during the usual care and closed-loop BG control portions of the study.
* History of eating disorder such as anorexia, bulimia, "diabulemia" or omission of insulin to manipulate weight
* History of intentional, inappropriate administration of insulin leading to severe hypoglycemia requiring treatment
* Any factors that, in the opinion of the principal investigator, would interfere with the safe completion of the study procedures.

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 32 (Actual)
Dates: Start 2013-04; Primary Completion 2013-08 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Russell, MD PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Russell SJ, El-Khatib FH, Sinha M, Magyar KL, McKeon K, Goergen LG, Balliro C, Hillard MA, Nathan DM, Damiano ER. Outpatient glycemic control with a bionic pancreas in type 1 diabetes. N Engl J Med. 2014 Jul 24;371(4):313-325. doi: 10.1056/NEJMoa1314474. Epub 2014 Jun 15. PMID 24931572
- See also: Information about this and related studies — http://www.bionicpancreas.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Bionic Pancreas Then Usual Care; Usual Care Then Bionic Pancreas: Subjects were campers or counselors between the ages of 12 and 21 years who had at least a 1-year history of type 1 diabetes mellitus and were receiving insulin pump therapy.
  In a random cross over design, subjects were assigned to either intervention (5 days on bionic pancreas) or standard care (5 days on insulin pump) with a 2 day washout period in between.
Period: Overall Study
Arm/Group | Bionic Pancreas Then Usual Care | Usual Care Then Bionic Pancreas
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Cross over design, 16 participants in each arm and then switched to second arm after a 1 day washout period.
Groups:
- All Study Participants: The bionic pancreas (closed loop) will be compared to usual care (subject's own insulin pump) in a crossover design in which each volunteer will serve as his or her own control. Each volunteer will be under closed-loop glucose control for five days and usual camp level of diabetes care for five days in random order with a two day washout period in between.
Arm/Group | All Study Participants
Number analyzed (Participants) | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 16 (3)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Total number of participants was 32. Half were allocated to each of the 2 arms and then switched to the other arm in a random cross over design so that data was obtained from each participant for each of the 2 arms.
  Participants
    All study participants: Female | 16
    All study participants: Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Difference in Average Blood Glucose (BG) Between Closed-loop (Bionic Pancreas Arm) and Open-loop (Insulin Pump Arm) Periods as Determined From All Scheduled HemoCue Measurements With Mean Evenly Weighted Across the Daytime and Nighttime Hours.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Bionic Pancreas | Control
Number analyzed (Participants) | 32 | 32
mg/dL | 138 (18) | 157 (27)

2. Primary Outcome: Percentage of Time With a Low Plasma Glucose Reading (Less Than 70mg/dl) in the Bionic Pancreas Arm as Compared to Insulin Pump Arm
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Bionic Pancreas | Standard Care (Insulin Pump)
Number analyzed (Participants) | 32 | 32
percentage of time | 6.1 (4.5) | 7.6 (7.3)

3. Secondary Outcome: Difference Between Closed-loop (Bionic Pancreas Arm) and Open-loop (Insulin Pump Arm) in Average BG as Determined From All HemoCue Measurements Taken During the Day/Nighttime Including All Extra Measurements.
Description: Difference between Closed-loop (Bionic Pancreas Arm) and Open-loop (Insulin Pump Arm) in average BG as determined from all HemoCue measurements taken during the day/nighttime including all extra measurements taken before meals, taken during exercise, and taken for hypoglycemia monitoring.
Time Frame: 1 week
Population: This data was not analysed to prevent bias. This information would have been misleading (unscheduled BG checks were performed to confirm a low BG mostly). Overall CGM trend, incidence/duration of hypoglycemia and BG trend during and after exercise is separately analyzed under other secondary outcomes.
Groups:
- Bionic Pancreas: Subjects were campers or counselors between the ages of 12 and 21 years who had at least a 1-year history of type 1 diabetes mellitus and were receiving insulin pump therapy.
  In a random cross over design, subjects were assigned to either intervention (5 days on bionic pancreas) or standard care (5 days on insulin pump) with a 1 day washout period in between.
Arm/Group | Bionic Pancreas
Number analyzed (Participants) | 0

4. Secondary Outcome: Difference Between Closed-loop (Bionic Pancreas Arm) and Open-loop (Insulin Pump Arm) in Number of Subjects With Mean BG < 154 mg/dl
Time Frame: Day 2-5
Measure: Count of Participants; unit: Participants
Arm/Group | Bi-hormonal Bionic Pancreas | Usual Care
Number analyzed (Participants) | 32 | 32
Participants | 29 | 14

5. Secondary Outcome: Difference in the Percentage of Study Days With Mean CGM BG </= 154 mg/dl Over the Duration of the Closed-loop Period vs. the Usual Care Period
Time Frame: Day 2-5
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Bi-hormonal Bionic Pancreas | Usual Care
Number analyzed (Participants) | 32 | 32
percentage of days | 75 (21.5) | 49.3 (36.2)

6. Secondary Outcome: Difference Between Closed-loop (Bionic Pancreas Arm) and Open-loop (Insulin Pump Arm) in Number of Hypoglycemic Events (BG <70mg/dl) as Determined From HemoCue Measurements
Time Frame: Day 1-5
Measure: Number; unit: events
Arm/Group | Bi-hormonal Bionic Pancreas | Usual Care
Number analyzed (Participants) | 32 | 32
events | 97 | 210

7. Secondary Outcome: Difference Between Closed-loop (Bionic Pancreas Arm) and Open-loop (Insulin Pump Arm) in Fraction of Time Spent Within CGMG (Continuous Glucose Monitor) Ranges (< 70 mg/dl, 70-120 mg/dl, 70-180 mg/dl, > 180 mg/dl, > 250 mg/dl)
Time Frame: 1 week
Population: Fraction of time < 70 mg/dl, 70-120 mg/dl, 70-180 mg/dl, > 180 mg/dl, > 250 mg/dl
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Bi-hormonal Bionic Pancreas | Usual Care
Number analyzed (Participants) | 32 | 32
percentage of time
  <70 mg/dl | 2.7 (2.2) | 5.3 (4.6)
  70-120 mg/dl | 39.4 (8.2) | 29.9 (12.3)
  70-180 mg/dl | 73.3 (9.0) | 63.8 (13.3)
  >180 mg/dl | 24.0 (8.5) | 30.9 (15.0)
  >250 mg/dl | 7.6 (5.6) | 10.8 (8.7)

8. Secondary Outcome: Difference Between Closed-loop (Bionic Pancreas Arm) and Open-loop (Insulin Pump Arm) in Mean BG During Exercise
Time Frame: 1 week
Population: Data on exercise not collected
Arm/Group | Bi-hormonal Bionic Pancreas | Usual Care
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Difference Between Closed-loop (Bionic Pancreas Arm) and Open-loop (Insulin Pump Arm) in Number of Severe Hypoglycemic Episodes and Nadir BG During Exercise
Time Frame: 1 week
Population: Individual data during exercise was not analyzed. No episodes of severe hypoglycemia were observed on bionic pancreas and only 1 episode of severe hypoglycemia occurred in usual care arm (insulin pump)
Measure: Count of Participants; unit: Participants
Arm/Group | Bi-hormonal Bionic Pancreas | Usual Care
Number analyzed (Participants) | 32 | 32
Participants | 0 | 1

10. Secondary Outcome: Difference in Mean CGMG on Day 1 vs. Remaining Days (Days 2-5) Between Closed Loop (Bionic Pancreas Arm) and Usual Care (Insulin Pump Arm)
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Bi-hormonal Bionic Pancreas | Usual Care
Number analyzed (Participants) | 32 | 32
mg/dl
  Mean CGMG on Day 1 | 169.2 (31.3) | 156 (37.0)
  Mean CGMG day 2-5 | 142 (12) | 158 (27)

11. Secondary Outcome: Difference Between Closed-loop (Bionic Pancreas) and Open-loop (Insulin Pump) in Mean Continuous Glucose Monitoring Glucose (CGMG)
Description: Day 2-5
Time Frame: Day 2-5
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Bionic Pancreas | Control
Number analyzed (Participants) | 32 | 32
mg/dl | 142 (12) | 158 (27)

12. Secondary Outcome: Difference Between Closed-loop and Open-loop in Area Over the Curve and Below 70 mg/dl (Measure of Total Hypoglycemia Exposure)
Time Frame: 1 week
Population: This outcome was not analyzed as we feel that the outcome "percentage of time <70mg/dl" is an equivalent indicator of hypoglycemia exposure instead of area over the curve, and can be used to compare outcomes with other studies.
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

13. Secondary Outcome: Difference Between Closed-loop (Bionic Pancreas Arm) and Open-loop (Insulin Pump Arm) in Area Over the Curve and Below 50 mg/dl (Measure of Total Hypoglycemia Exposure)
Time Frame: 1 week
Population: This outcome was not analyzed as we feel that the outcome "percentage of time <50mg/dl" is a n equivalent indicator of severe hypoglycemia instead of area over the curve, and can be used to compare outcomes with other studies.
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

14. Secondary Outcome: Difference Between Closed-loop (Bionic Pancreas Arm) and Open-loop (Insulin Pump Arm) in Number of Subjects With Mean CGMG < 154 mg/dl
Time Frame: 1 week
Measure: Count of Participants; unit: Participants
Arm/Group | Bi-hormonal Bionic Pancreas | Usual Care
Number analyzed (Participants) | 32 | 32
Participants | 26 | 17

15. Secondary Outcome: Difference Between Closed-loop and Open-loop in Mean CGMG in the Four Hour Period Following Meals
Time Frame: 1 week
Population: Data was not collected to measure this outcome
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

16. Secondary Outcome: Difference Between Closed-loop (Bionic Pancreas Arm) and Open-loop (Insulin Pump Arm) in Mean CGMG During Exercise
Time Frame: 1 week
Population: Data not obtained for exercise period
Arm/Group | Bi-hormonal Bionic Pancreas | Usual Care
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Difference Between Closed-loop (Bionic Pancreas Arm) and Open-loop (Insulin Pump Arm) in Standard Deviation of CGMG Values (Glycemic Variability) in Different BG Ranges.
Description: Difference between Closed-loop (Bionic Pancreas Arm) and Open-loop (Insulin Pump Arm) in standard deviation of CGMG values (glycemic variability) in different BG ranges.
  %<70 70-120 70-180 %>180 %>250
Time Frame: 1 week
Measure: Number; unit: Standard deviation of mean values
Arm/Group | Bi-hormonal Bionic Pancreas | Usual Care
Number analyzed (Participants) | 32 | 32
Standard deviation of mean values
  <70 | 2.2 | 4.6
  70-120 | 8.2 | 12.3
  70-180 | 9.0 | 13.3
  >180 | 8.5 | 15.0
  >250 | 5.6 | 8.7

18. Secondary Outcome: Difference Between Closed-loop (Bionic Pancreas Arm) and Open-loop (Insulin Pump Arm) in Standard Deviation of CGMG Values at Night (11:00 PM to 7:00 AM)
Time Frame: 1 week
Measure: Number; unit: Standard deviation of mean values
Arm/Group | Bi-hormonal Bionic Pancreas | Usual Care
Number analyzed (Participants) | 32 | 32
Standard deviation of mean values
  <70 | 2.1 | 5.4
  70-120 | 12.3 | 17.1
  70-180 | 8.5 | 16.9
  >180 | 7.6 | 19.8
  >250 | 3.4 | 10.9

19. Secondary Outcome: Difference Between Closed-loop and Open-loop in Average BG as Determined From All HemoCue Measurements Taken During the Nighttime Including All Extra Measurements Taken for Hypoglycemia Monitoring.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Bi-hormonal Bionic Pancreas | Usual Care
Number analyzed (Participants) | 32 | 32
mg/dl | 141 (20) | 162 (37)

20. Secondary Outcome: Difference Between Closed-loop (Bionic Pancreas Arm) and Open-loop (Insulin Pump Arm) in Time Spent in Hypoglycemia (Plasma BG <Than 70 mg/dl) at Night
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Bi-hormonal Bionic Pancreas | Usual Care
Number analyzed (Participants) | 32 | 32
percentage of time | 4.1 (6.1) | 4.4 (6.7)

21. Secondary Outcome: Difference Between Closed-loop and Open-loop in Fraction of Time at Night Spent Within Glucose Ranges (< 70 mg/dl, 70-120 mg/dl, 70-180 mg/dl, > 180 mg/dl, > 250 mg/dl)
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Bi-hormonal Bionic Pancreas | Usual Care
Number analyzed (Participants) | 32 | 32
percentage of time
  <70 | 2.4 (2.1) | 5.0 (5.4)
  70-120 | 51.5 (12.3) | 27.4 (17.1)
  70-180 | 84.6 (8.5) | 65.9 (16.9)
  >180 | 13.0 (7.6) | 29.8 (19.8)
  >250 | 2.8 (3.4) | 8.6 (10.9)

22. Secondary Outcome: Difference Between Closed-loop (Bionic Pancreas Arm) and Open-loop (Insulin Pump Arm) in Mean CGMG at Night
Description: Day 2-5
Time Frame: Day 2-5
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Bionic Pancreas | Control
Number analyzed (Participants) | 32 | 32
mg/dl | 124 (11) | 157 (36)

23. Secondary Outcome: Difference Between Closed-loop (Bionic Pancreas Arm) and Open-loop (Insulin Pump Arm) in Fraction of Time Spent Within CGMG Ranges (< 70 mg/dl, 70-120 mg/dl, 70-180 mg/dl, > 180 mg/dl, > 250 mg/dl) at Night
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Bionic Pancreas | Control
Number analyzed (Participants) | 32 | 32
percentage of time
  <70 mg/dl | 2.6 (2.5) | 4.0 (5.3)
  70-120 mg/dl | 55.3 (13.7) | 28.3 (17.3)
  70-180 mg/dl | 86.9 (8.1) | 66.7 (19.9)
  >180 mg/dl | 10.5 (7.0) | 29.3 (22.0)
  >250 mg/dl | 1.8 (2.5) | 9.5 (12.5)

24. Secondary Outcome: Difference Between Closed-loop and Open-loop in Area Over the Curve and Below 70 mg/dl (Measure of Total Hypoglycemia Exposure) at Night
Time Frame: 1 week
Population: This outcome was not analyzed as we feel that the outcome "percentage of time <70mg/dl at nightime" is an equivalent indicator of overnight hypoglycemia exposure instead of area over the curve, and can be used to compare outcomes with other studies.
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

25. Secondary Outcome: Difference Between Closed-loop and Open-loop in Area Over the Curve and Below 50 mg/dl (Measure of Total Hypoglycemia Exposure) at Night
Time Frame: 1 week
Population: This outcome was not analyzed as we feel that the outcome "percentage of time <50mg/dl at nightime" is an equivalent indicator of severe overnight hypoglycemia exposure instead of area over the curve, and can be used to compare outcomes with other studies.
Arm/Group | All Study Participants
Number analyzed (Participants) | 0

26. Secondary Outcome: Difference Between Closed-loop (Bionic Pancreas Arm) and Open-loop (Insulin Pump Arm) in Number of Carbohydrate Interventions for Hypoglycemia
Time Frame: 1 week
Measure: Number; unit: number of interventions
Arm/Group | Bionic Pancreas | Control
Number analyzed (Participants) | 32 | 32
number of interventions | 97 | 210

27. Secondary Outcome: Difference Between Closed-loop (Bionic Pancreas Arm) and Open-loop (Insulin Pump Arm) in Number of Carbohydrate Interventions for Hypoglycemia at Night
Time Frame: 1 week
Measure: Number; unit: interventions
Arm/Group | Bionic Pancreas | Control
Number analyzed (Participants) | 32 | 32
interventions | 29 | 48

28. Other Pre Specified Outcome: Difference Between Closed-loop (Bionic Pancreas Arm) and Open-loop (Insulin Pump Arm) in Mean Insulin Total Daily Dose
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: unit/kg/day
Arm/Group | Bionic Pancreas | Control
Number analyzed (Participants) | 32 | 32
unit/kg/day | 0.82 (0.16) | 0.79 (0.17)

ADVERSE EVENTS:
Arm/Group | Bionic Pancreas | Control
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 6/32 | 4/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bionic Pancreas (N=32) | Control (N=32)
Episodes of Severe Hypoglycemia (Endocrine disorders) | 0 | 1
Transient hyperketonemia (Endocrine disorders) | 3 | 3
Nausea (Endocrine disorders) | 1 | 0
Vomiting (Endocrine disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-02-12): https://cdn.clinicaltrials.gov/large-docs/88/NCT01833988/Prot_SAP_001.pdf